CLINICAL TRIAL: NCT01035697
Title: A Study to Determine If Inflammatory Cytokines Are Associated With Perinatal Brain Injury and Long Term Neurodevelopmental Handicap or Death
Brief Title: Inflammatory Cytokines Associated With Perinatal Brain Injury
Acronym: Cytokines
Status: Completed | Type: Observational
Sponsor: NICHD Neonatal Research Network (Network)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency); National Center for Research Resources (NCRR) (NIH)
Responsible Party: Waldemar A. Carlo, MD, Lead Principal Investigator, University of Alabama at Birmingham
Other Study IDs: NICHD-NRN-0022; U10HD027853 (NIH); M01RR008084 (NIH); U10HD040492 (NIH); M01RR000030 (NIH); U10HD027851 (NIH); M01RR000039 (NIH); U10HD027856 (NIH); M01RR000750 (NIH); U10HD021364 (NIH); M01RR000080 (NIH); U01HD036790 (NIH); U10HD027880 (NIH); M01RR000070 (NIH); U10HD034216 (NIH); M01RR000032 (NIH); U10HD040461 (NIH); U10HD021397 (NIH); M01RR016587 (NIH); U10HD027881 (NIH); M01RR000997 (NIH); U10HD021415 (NIH); U10HD040689 (NIH); M01RR000633 (NIH); U10HD021373 (NIH); U10HD040498 (NIH); M01RR007122 (NIH); U10HD021385 (NIH); U10HD027904 (NIH); U10HD027871 (NIH); M01RR006022 (NIH)
Record Dates: First submitted 2009-12-17; First posted 2009-12-21 (Estimated); Last update posted 2019-03-22 (Actual); Status verified 2019-03

CONDITIONS: Infant, Newborn; Infant, Low Birth Weight; Infant, Small for Gestational Age; Infant, Premature; Cerebral Palsy
Keywords: NICHD Neonatal Research Network; Very Low Birth Weight (VLBW); Extremely Low Birth Weight (ELBW); Prematurity; Pro-inflammatory cytokines; Anti-inflammatory cytokines; Interleukin-1 (IL-1β); Interleukin-2 (IL-2); Interleukin-3 (IL-3); Interleukin-8 (IL-8); Interleukin-9 (IL-9); Tumor necrosis factor-α (TNF-α); Regulated upon Activation, Normal T-cell Expressed and Secreted (RANTES)
MeSH Terms: conditions — Premature Birth; Cerebral Palsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood spots collected on filter paper.
Oversight: Data Monitoring Committee: No

SUMMARY:
This observational study assessed whether measurements of certain pro-inflammatory and anti-inflammatory cytokines in the blood (either singly or in combination) at birth and/or up to day of life 21 can predict cerebral palsy at 18-22 months corrected age.

DETAILED DESCRIPTION:
Inflammatory cytokines [interleukin-1 (IL-1β), IL-8, IL-9, tumor necrosis factor-α (TNF-α), and RANTES] but not anti-inflammatory cytokines released during the perinatal period have been associated with the development of periventricular leukomalacia (PVL) and cerebral palsy (CP) in near term and term infants. However, because blood samples were obtained on any day between day 1 and 18, these data cannot distinguish between prenatal and postnatal effects on neurological outcome. Furthermore, very low birth weight infants who are at the highest risk have not been studies.

The goal of this study was to measure pro-inflammatory and anti-inflammatory cytokine levels at various times in the perinatal period (at birth up to day of life 21), since they may be elevated at different points in the disease process. Blood samples (whole blood spots, dried on filter paper) were obtained on day 1 within 4 hours after birth, and on days 3, 7, 14, and 21. Neurodevelopmental assessments were conducted at 18-22 months corrected age.

ELIGIBILITY:
Inclusion Criteria:

* Infants 401-1,000 grams at birth

Exclusion Criteria:

* >72 hours of age

Max Age: 72 Hours | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Infants 401-1,000 grams at birth of both genders and all racial/ethnic groups.
Sampling Method: Probability Sample
Enrollment: 1067 (Actual)
Dates: Start 1999-07; Primary Completion 2002-07 (Actual); Study Completion 2004-05 (Actual)

PRIMARY OUTCOMES:
Pro-cytokines increased and anti-inflammatory cytokines decreased | At birth and/or up to Day 3±1

SECONDARY OUTCOMES:
Type and severity of CP and other neurodevelopmental handicaps, the appearance of PVL, and neonatal mortality | 18-22 months corrected age
Abnormal pro-inflammatory and anti-inflammatory cytokines at birth are associated with prenatal insults (e.g., chorioamnionitis, occult intrauterine infection, early-onset neonatal sepsis, perinatal asphyxia, early death) | At birth
Abnormal postnatal cytokine levels associated with postnatal insults (e.g., postnatal intraventricular hemorrhage, late-onset neonatal sepsis, bronchopulmonary dysplasia, chronic lung disease, and/or necrotizing enterocolitis) | Up to Day of life 21
Pro-inflammatory cytokine elevations at the time of a workup for possible sepsis occur in infants with a positive bacterial blood culture and those with negative blood cultures who are treated with a full course of antibiotics | Up to Day of life 21

CONTACTS AND LOCATIONS:
Overall Officials: William Oh, MD, Principal Investigator — Brown University, Women & Infants Hospital of Rhode Island; Michele C. Walsh, MD MS, Principal Investigator — Case Western Reserve University, Rainbow Babies & Children's Hospital; Ronald N. Goldberg, MD, Principal Investigator — Duke University; Barbara J. Stoll, MD, Principal Investigator — Emory University; James A. Lemons, MD, Principal Investigator — Indiana University; Abhik Das, PhD, Principal Investigator — RTI International; David K. Stevenson, MD, Principal Investigator — Stanford University; Waldemar A. Carlo, MD, Principal Investigator — University of Alabama at Birmingham; Neil N. Finer, MD, Principal Investigator — University of California, San Diego; Edward F. Donovan, MD, Principal Investigator — Children's Hospital Medical Center, Cincinnati; Shahnaz Duara, MD, Principal Investigator — University of Miami; Lu-Ann Papile, MD, Principal Investigator — University of New Mexico; Sheldon B. Korones, MD, Principal Investigator — University of Tennessee; Jon E. Tyson, MD MPH, Principal Investigator — The University of Texas Health Science Center, Houston; Abbot R. Laptook, MD, Principal Investigator — University of Texas; T. Michael O'Shea, MD MPH, Principal Investigator — Wake Forest University; Seetha Shankaran, MD, Principal Investigator — Wayne State University; Richard A. Ehrenkranz, MD, Principal Investigator — Yale University
Locations (18):
- United States (18):
  - University of Alabama, Birmingham, Alabama
  - Stanford University, Palo Alto, California
  - University of California at San Diego, San Diego, California
  - Yale University, New Haven, Connecticut
  - University of Miami, Miami, Florida
  - Emory University, Atlanta, Georgia
  - Indiana University, Indianapolis, Indiana
  - Wayne State University, Detroit, Michigan
  - University of New Mexico, Albuquerque, New Mexico
  - Wake Forest University, Charlotte, North Carolina
  - RTI International, Durham, North Carolina
  - Duke University, Durham, North Carolina
  - Cincinnati Children's Medical Center, Cincinnati, Ohio
  - Case Western Reserve University, Rainbow Babies and Children's Hospital, Cleveland, Ohio
  - Brown University, Women & Infants Hospital of Rhode Island, Providence, Rhode Island
  - University of Tennessee, Memphis, Tennessee
  - University of Texas Southwestern Medical Center at Dallas, Dallas, Texas
  - University of Texas Health Science Center at Houston, Houston, Texas

REFERENCES:
- [Result] Ambalavanan N, Carlo WA, D'Angio CT, McDonald SA, Das A, Schendel D, Thorsen P, Higgins RD; Eunice Kennedy Shriver National Institute of Child Health and Human Development Neonatal Research Network. Cytokines associated with bronchopulmonary dysplasia or death in extremely low birth weight infants. Pediatrics. 2009 Apr;123(4):1132-41. doi: 10.1542/peds.2008-0526. PMID 19336372
- [Result] Natarajan G, Shankaran S, McDonald SA, DAS A, Stoll BJ, Higgins RD, Thorsen P, Skogstrand K, Hougaard DM, Carlo WA; NICHD neonatal research network. Circulating beta chemokine and MMP 9 as markers of oxidative injury in extremely low birth weight infants. Pediatr Res. 2010 Jan;67(1):77-82. doi: 10.1203/PDR.0b013e3181c0b16c. PMID 19755933
- [Result] Sood BG, Madan A, Saha S, Schendel D, Thorsen P, Skogstrand K, Hougaard D, Shankaran S, Carlo W; NICHD neonatal research network. Perinatal systemic inflammatory response syndrome and retinopathy of prematurity. Pediatr Res. 2010 Apr;67(4):394-400. doi: 10.1203/PDR.0b013e3181d01a36. PMID 20032809
- [Result] Carlo WA, McDonald SA, Tyson JE, Stoll BJ, Ehrenkranz RA, Shankaran S, Goldberg RN, Das A, Schendel D, Thorsen P, Skogstrand K, Hougaard DM, Oh W, Laptook AR, Duara S, Fanaroff AA, Donovan EF, Korones SB, Stevenson DK, Papile LA, Finer NN, O'Shea TM, Poindexter BB, Wright LL, Ambalavanan N, Higgins RD; Eunice Kennedy Shriver National Institute of Child Health and Human Development Neonatal Research Network. Cytokines and neurodevelopmental outcomes in extremely low birth weight infants. J Pediatr. 2011 Dec;159(6):919-25.e3. doi: 10.1016/j.jpeds.2011.05.042. Epub 2011 Jul 27. PMID 21798559
- See also: NICHD Neonatal Research Network — http://neonatal.rti.org/